CLINICAL TRIAL: NCT06302933
Title: Negative Serology by Immunoenzymatic Test (EIA) in HIV-infected Children Treated Early With Antiretroviral in the ANRS-Pediacam Study: Pathophysiological Mechanisms
Acronym: PediacamNEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Centre Pasteur du Cameroun (Other); Centre Mère et Enfant de la Fondation Chantal Biya (Other); Centre Hospitalier D'essos (Other); Hospital General De Douala (Other); CH Orléans (Unknown); Institut Pasteur (Industry); Hopital Universitaire Robert-Debre (Other); Université Paris-Sud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ANRS 12414 PediacamNEG
Record Dates: First submitted 2023-08-24; First posted 2024-03-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Study type: a study nested in the ANRS 12225 - Pediacam III cohort, comprising two phases
  * A retrospective phase: case-control study The analyzed data are those collected previously or measured from the already available bio bank, within the framework of the Pediacam III cohort during the primary infection phase before the initiation of HAART, at 6 months after the end of the first series of EPI vaccines, and at 2 years.
  * A prospective phase: cross-sectional study Based on an ad hoc bio bank created for parameters we couldn't measure on the existing bio bank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children enrolled in Pediacam III ANRS12225 cohort (Other)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood samples collected from children followed in the Pediacam III ANRS12225 cohort

SUMMARY:
The objective of the study is to identify the pathophysiological mechanisms responsible for the induction and maintenance of negative serologies by EIA tests in HIV-infected children treated early with HAART in the ANRS 12225-Pediacam III cohort in Cameroon

The hypothesis of better control of HIV infection through interactions between immunological, viral, and genetic factors was made to build the following objectives:

* Immunological aspect: lack of humoral response or immune activation
* Virological aspect: Reduced HIV reservoir size
* Determine the HLA phenotype in the different groups of children included and the KIR genotypes.

DETAILED DESCRIPTION:
There will be two phases of the study :

* A retrospective phase: case-control study The analyzed data are those collected previously or measured from the already available bio bank, within the framework of the Pediacam III cohort during the primary infection phase before the initiation of HAART, at 6 months after the end of the first series of EPI vaccines, and at 2 years.
* A prospective phase: cross-sectional study Based on an ad hoc bio bank created for parameters we couldn't measure on the existing bio bank

ELIGIBILITY:
Inclusion Criteria:

Case control study

* Children included and followed in the ANRS 12225 study - Pediacam III
* Having plasma samples in the bio bank during the above-mentioned periods Case:children with at least one negative HIV serology made by ELISA, permanent or transientduring follow-up.

Control (4 groups)

* HIV-infected children with positive serology and viral load (VL) <400 copies /ml
* HIV-infected children with positive serology and VL ≥400 copies / ml
* HIV-uninfected children born to HIV-positive mothers
* HIV-uninfected children born to HIV-uninfected mothers Selection of cases and controls will be matched on gestational age (premature <37, term ≥37 weeks) and year of birth (2007-2008 and 2009-2010).

Cross sectional study Inclusion criteria

* All children still followed in the ANRS - Pediacam III cohort
* Written consent of one of the parents or the guardian and assent of the child if aged ≥ 11 years and complete disclosure of HIV statusfor infected children for participation to the study.

Exclusion Criteria:

* Refusal by one of the parents or the guardian for the child's participation in the study
* No assent of the child (if aged ≥ 11 years and with complete disclosure of HIV status, for infected children)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of sCD14 (µg/ml). Levels of these biomarkers will be compared across all groups.
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of BAFF using luminex or commercially available ELISA quantification kits. Levels of these biomarkers will be compared across all groups.
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of CXCL13 using luminex or commercially available ELISA quantification kits. Levels of these biomarkers will be compared across all groups.
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of TNF-α (pg/ml). Levels of these biomarkers will be compared across all groups.
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of IL-10 (pg/ml). Levels of these biomarkers will be compared across all groups.
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of IP-10 (pg/ml). Levels of these biomarkers will be compared across all groups.
Level of pro-inflammatory and anti-inflammatory cytokines, chimiokines in the plasma | 18 months
  Measure of TRAIL (ng/ml). Levels of these biomarkers will be compared across all groups

SECONDARY OUTCOMES:
- Humoral response to vaccines against tetanus, pertussis, and viral hepatitis B | 18 months
  Serum concentrations of human IgG antibodies against tetanus-toxoid, pertussis, and viral hepatitis B will be measured using commercially available ELISA quantification kits and results will be given as IU/mL
- Functional and phenotypic characterization of B and T lymphocytes | 18 months
  Level (cells/μL or percentage) of T and B-cell lymphocytes subpopulations will be assess in blood using flow cytometry. Functional characterization of T and B lymphocytes will be done by cell culture following by cytokine production titration
- Size of the HIV reservoir | 18 months
  Measure total (copies/million PBMC), integrated (copies/million PBMC), unintegrated (copies/million PBMC) HIV DNA level in Peripheral Blood Mononuclear Cells (PBMC)
- Residual viremia in perinatally HIV-infected adolescent | 18 months
  Any detectable HIV-RNA below 50 copies/mL
- Level of HIV plasma p24 | 18 months
  Measure plasma level of HIV p24 antigen (fg/ml) using ultrasentsitive technique called Simoa (Single molecule array)
- HLA phenotype and the KIR genotypes | 18 months
  HLA-B (27 et 57), HLA-B35 ou 53, HLA-C16:01+KIR2DL3+

CONTACTS AND LOCATIONS:
Locations (3):
- Cameroon (3):
  - Hôpital de Jour - Hôpital Laquintinie de Douala, Douala
  - Unité Pédiatrique de Jour - Centre Mère et Enfant de la Fondation Chantal Biya, Yaoundé
  - Service de Pédiatrie - Centre Hospitalier d'Essos, Yaoundé